CLINICAL TRIAL: NCT02167386
Title: PrEP for Black MSM: Community-Based Ethnography and Clinic-Based Treatment
Brief Title: PrEPared and Strong: Clinic-Based PrEP for Black MSM
Acronym: P&S
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Columbia University (Other)
Collaborators: National Institute of Mental Health (NIMH) (NIH); Gilead Sciences (Industry)
Responsible Party: Principal Investigator, Paul Colson, Associate Research Scientist, Columbia University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: AAAO0852; 5R01MH098723 (NIH)
Record Dates: First submitted 2014-06-12; First posted 2014-06-19 (Estimated); Last update posted 2018-05-17 (Actual); Status verified 2018-05

CONDITIONS: HIV/AIDS
Keywords: Men who have sex with men (MSM); Black/African-American
MeSH Terms: conditions — Acquired Immunodeficiency Syndrome; Homosexuality

STUDY DESIGN:
Intervention Model Description: combination drug and behavioral intervention
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Enhanced PrEP Adherence (Experimental): Enhanced PrEP Adherence: peer navigators, PrEP support group, on-line support group, text message reminders
  Interventions: Behavioral: Enhanced PrEP Adherence
- Standard PrEP Adherence (Active Comparator): Standard PrEP Adherence: support groups, case management
  Interventions: Behavioral: Standard PrEP Adherence

INTERVENTIONS:
Behavioral: Enhanced PrEP Adherence
  Arms: Enhanced PrEP Adherence
Behavioral: Standard PrEP Adherence
  Arms: Standard PrEP Adherence

SUMMARY:
Black men who have sex with men (MSM) have among the highest rates of new HIV infections of any group in the United States. Developing effective HIV prevention interventions that work with this group is a critical element of the National HIV/AIDS Strategy. In the first phase of our study ("the ethnographic phase"), the investigators will carry out community-based research that will explore structural, social and cultural factors relevant to how Black MSM might engage with Pre-Exposure Prophylaxis (PrEP). This phase of community-based research will inform the design of an enhanced PrEP adherence intervention, which will be subsequently tested at a community-based health clinic in Harlem in the second phase of the project.

DETAILED DESCRIPTION:
STUDY OBJECTIVES AND DESIGN This randomized clinical trial will enroll HIV-uninfected Black MSM and transgender females (TGF) and randomly assign them to receive enhanced versus standard PrEP adherence packages. Study participants will receive PrEP-related clinical care at Harlem United, a community-based healthcare provider in New York City's Central Harlem.

Primary Objective Compare the effectiveness of enhanced versus standard packages for increasing adherence to PrEP in a community-based primary care clinic

Secondary Objectives

1. Compare the enhanced and standard PrEP adherence packages on:

   * sexual risk behaviors
   * retention in care
   * PrEP knowledge
   * seroconversions
2. Examine the safety of PrEP among participants as measured by the type and frequency of adverse events
3. Describe acceptability of daily PrEP among Black MSM and TGF generally and among those who have agreed to take PrEP

Study Design This is an open-label, randomized clinical trial that aims to assess the effectiveness of an enhanced PrEP adherence package compared to a standard PrEP adherence package on PrEP adherence. PrEP uptake, acceptability, safety, retention in care, and feasibility will also be measured. Participants will be prescribed once daily oral co-formulated emtricitabine/tenofovir disoproxil fumarate (Truvada) by physicians at Harlem United, a community-based primary-care clinic located in Harlem, New York City. 200 participants will be recruited through: Harlem United client services; studies being conducted at the Harlem Prevention Center; the study's ethnographic component; and targeted direct recruitment strategies. Each participant will receive PrEP for one year. In addition to PrEP, all participants will receive comprehensive HIV prevention services with access to condoms, risk reduction counseling, and STI screening and treatment. Participants will have follow up clinical visits at 12 week intervals to be evaluated for side effects, renal toxicity, adherence, risk behavior, and HIV seroconversion.

Additionally, the study will assess: 1) correlates of PrEP knowledge, uptake, safety, retention in care, and acceptability among Black MSM and TGF individuals who are determined to be eligible for PrEP based on self-reported sexual risk behavior and history of sexually transmitted infections (STIs); and 2) patterns and correlates of adherence among participants in the study. The project will also assess other aspects of PrEP feasibility including risk compensation and side effects.

The first eligible 50 individuals who are agree to be in the study but decline to take PrEP will be asked to answer a brief set of questions about the reasons for their decision.

STUDY POPULATION

Description of Study Site The study will be implemented in Harlem, New York by the Harlem Prevention Center (HPC), Mailman School of Public Health, Columbia University. HPC is located on 125th Street in Central Harlem and is the home for various HIV and tuberculosis (TB) studies, including HIV prevention studies. Informed consent and research interviews will be conducted and study records stored at HPC.

Harlem United (HU), a community-based organization offering health and social services in Central Harlem, will serve as the locus of many study activities. HU has the capacity to comply with the protocol, project-specific procedures, and all applicable regulations. HU locations include 1) HOME (Helping Our Members Evolve), a drop-in center for younger MSM and TGF clients, 2) the Prevention Center which provides non-clinical HIV and non-HIV services to clients of all ages and genders, and 3) the Willis P. Green Jr Clinic providing HIV and non-HIV medical services. All sites have reception areas with waiting areas, counseling rooms, private rooms for HIV testing, and data management areas. Additionally, the clinic has physical examination rooms, medication storage areas, and access to laboratory facilities.

Description of Study Population The study population is Black MSM and TGF, who are at-risk for HIV infection. MSM and TGF at-risk for HIV infection are defined as men or male-to-female transgendered individuals who report indicators of HIV risk. We expect that approximately 95% of participants will be MSM due to their larger population size in the Harlem community.

STUDY PROCEDURES Individuals who meet criteria for the study will receive a referral for medical assessment. Individuals who are medically eligible to take PrEP and who agree to initiate PrEP will provide Informed Consent. They will then be given a 30-day PrEP prescription, followed by a baseline research interview. After enrollment, participants will be seen for a 4-week follow-up visit to be evaluated for evidence of HIV seroconversion, adherence to medication, and clinical toxicity. Subsequent medical and research follow-up visits will occur at 3, 6, 9, and 12 months after enrollment. Quarterly medical visits will include testing for HIV and STIs as per clinic protocol. In addition, study participants will have creatinine levels checked and will receive brief adherence and risk reduction counseling. Participants who wish to discontinue PrEP will remain in the study and may resume PrEP. Those who discontinue PrEP and wish to leave the study will be asked to complete an exit interview.

ELIGIBILITY:
Inclusion Criteria:

* male at birth
* self-identify as Black, African American, Caribbean Black, African, or multiethnic Black
* are 18 years of age or older
* any male or transgender woman (TGW) partners in past 6 months;
* not in a monogamous partnership with a recently tested, HIV-negative man;
* have at least one of the following:
* reporting condomless anal and/or receptive neovaginal intercourse with at least one man or TGW in the past six months;
* any STI diagnosed or reported in past 6 months;
* is in on-going sexual relationship with an HIV-positive male or TGW partner;
* able to provide written informed consent in English;
* able to provide a street address or residence or phone number for themselves or two personal contacts who would know their whereabouts during participation in the study

Exclusion Criteria:

* current participation in any other PrEP study;
* having taken PrEP in programmatic context more than 3 months

Min Age: 18 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 204 (Actual)
Dates: Start 2015-03-30 (Actual); Primary Completion 2018-02-28 (Actual); Study Completion 2018-02-28 (Actual)

PRIMARY OUTCOMES:
adherence to daily Truvada use | twelve months after enrollment
  this is a measure of PrEP adherence, to be implemented through self-reported adherence and collection of dried blood spots

SECONDARY OUTCOMES:
percentage of sexual acts where condom was used | twelve months after enrollment
  this is one measure of sexual risk behaviors. Other such measures include number and type of sexual partner, specific sexual acts, drug/alcohol use during sex, transactional sex
number of correct knowledge items | twelve months after enrollment
  this is one outcome measure from a knowledge, attitudes, and practices (KAP) questionnaire related to HIV prevention in general and PrEP in particular
number of participants remaining in care | end of 12-month study period
  this is a measure of retention in care. As each participants finishes his 12-month study period, retention will be determined by number of care visits completed.
positive HIV test | during 12-month study period
  this is a measure of seroconversion. Participants who test HIV-positive at any quarterly care visit will exit the study and will be referred for HIV care.

CONTACTS AND LOCATIONS:
Overall Officials: Paul W Colson, PhD, Principal Investigator — ICAP, Mailman School of Public Health, Columbia University
Locations (2):
- United States (2):
  - Harlem Prevention Center, New York, New York
  - Harlem United, New York, New York

REFERENCES:
- [Derived] Colson PW, Franks J, Wu Y, Winterhalter FS, Knox J, Ortega H, El-Sadr WM, Hirsch-Moverman Y. Adherence to Pre-exposure Prophylaxis in Black Men Who Have Sex with Men and Transgender Women in a Community Setting in Harlem, NY. AIDS Behav. 2020 Dec;24(12):3436-3455. doi: 10.1007/s10461-020-02901-6. PMID 32385678